CLINICAL TRIAL: NCT02411838
Title: A Pilot Study of Adipokines and Calorie Restriction in Multiple Sclerosis Patients
Brief Title: Calorie Restriction in Multiple Sclerosis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Laura Piccio, Research Assistamt Professor, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 201307106
Record Dates: First submitted 2013-12-05; First posted 2015-04-08 (Estimated); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; calorie restriction; adipokines
MeSH Terms: conditions — Multiple Sclerosis | interventions — Caloric Restriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): Steroid treatment (10 total days), which is a standard therapy for significant MS relapses.
- Calorie restriction (Experimental): The intervention in this group will be to undergo a regimen of calorie restriction through fasting every other day (named "alternate day fasting").
  Specifically this group will undergo alternate day fasting plus the same steroid regimen as the control group (CR GROUP).
  During the day of fasting the subject will be allowed to eat two salads with light dressing, not to go over approximately 500 calories. The CR group subjects will fast on day 2 (second day of IVMP) and then continue to fast on alternate days until day 15. This is the end of the Acute CR phase of the Study, and patients may discontinue the study at this point.
  Interventions: Other: Calorie restriction

INTERVENTIONS:
Other: Calorie restriction — Calorie restriction will be achieved by alternate day fasting. During the day of fasting the subject will be allowed to eat two salads with light dressing, not to go over approximately 500 calories. The CR group subjects will fast on day 2 (second day of steroids) and then continue to fast on alternate days until day 15. This is the end of the Acute CR phase of the Study, and patients may discontinue the study at this point.
  Chronic CR phase At the end of the Acute CR phase, both groups will be offered to enroll in the alternate day fasting regimen for 6 months (Chronic CR phase). During this phase, patients with a BMI <28 will follow a regimen of fasting for two days per week while patients with BMI>28 will follow a regimen of fasting for three days per week.
  Arms: Calorie restriction

SUMMARY:
The investigators hypothesize that adipokine (soluble molecules produced by the adipose tissue) levels are altered in MS compared to control subjects. Additionally, the investigators hypothesize that calorie restriction (CR) will improve clinical recovery from an MS relapse, ameliorate the adipokine and metabolic-inflammatory profile in MS, and enhance immune-regulatory mechanisms.

This is a pilot study to determine the effects of CR in MS patients during an acute MS relapse (Acute CR phase) and for 6 months afterwards (Chronic CR phase). Calorie restriction will be achieved by following a regimen of alternate day fasting. The investigators will evaluate clinical outcomes and blood biomarkers at different time points.

DETAILED DESCRIPTION:
The goal of this study is to determine the effects of CR on blood biomarkers (including serum levels of adipokines, cytokines, cortisol and T reg numbers) compared to standard therapies in MS patients during recovery from a relapse. Sixteen MS patients (body mass index-BMI ≥ 23) having an attack will be enrolled and randomized to either:

1. steroid treatment (10 days) which is standard therapy for MS relapses; or
2. CR plus steroid treatment (10 days). Calorie restriction will be achieved by following a regimen of alternate day fasting (during the day of fasting the subject will be allowed to eat two salads with olive oil and lemon juice or vinegar). Briefly, the subjects will fast on day 1 (first day of steroids) and then continue to fast on alternate days until day 15, another fasting day. After 15 days of alternate day fasting, both groups will be offered to enroll in the intermittent fasting regimen for 6 months (with salads allowed on the fasting day) (chronic CR phase). Specifically, patients with a BMI <28 will follow a regimen of fasting for two days per week while patients with BMI>28 will follow a regimen of fasting for three days per week. Blood samples will be obtained and analyzed at specified points during the study for routine testing (CBC and CMP) and immune/inflammatory analyses. Specifically, a blood sample will be obtained at baseline (day 1, before starting steroids) and after 15 days on alternate fasting. For those patients that will be enrolled in the chronic CR study for six months blood samples will also be obtained at month 3 and 6. MS subjects will be evaluated on day 15 after initiation of steroids. Those subjects that will participate in the chronic CR study will also donate blood at months 3 and 6. If patients are taking an immunomodulatory medication for MS, they will continue during the entire trial. They will be followed and assessed during the study by a nutritionist experienced with human CR. Patients will be seen by the nutritionist at baseline, day 15 for the first portion of the study. At the baseline visit they will be instructed to fast on day 1 and then every other day. During the fasting days, patients are allowed to eat a salad with 2 Table spoons of olive oil or canola oil plus vinegar or lemon juice twice/day. The goal is to eat less than 500 calories on fasting days. The nutritionist will also educate the patient to consume a nutritionally adequate diet during non-fasting days to avoid "overeating". Patients will keep a daily food diary and those entering the chronic CR phase will return to the center to meet with the nutritionist at months 3 and 6 (with telephone contacts in between).

At the baseline visit, patients will sign the informed consent, and the investigators will collect medical history, perform physical examination, calculate BMI (defined as weight in Kg / height in m2) and waist circumference (index of visceral fat accumulation) and perform neurological assessments, including the EDSS which is the standard neurologic exam used in MS trials which assigns a score from 0 (no deficit) to 10 (dead from MS), the multiple sclerosis functional composite (MSFC), which is a quantitative test of upper and lower limb function and cognition supplemented with an additional cognitive test called the Symbol Digit Modality Test (SDMT) and MS quality of life inventory (MSQLI).

Blood will be collected for routine testing (CBC, CMP) and for adipokine/cytokine, cortisol, and T reg cell analyses performed by the investigators' laboratory. All these assessments and sample collections will be repeated at day 15 and at month 3 and 6 for patients that will participate in the chronic CR phase. Neurologic exams will be also performed on day 2, 3 during steroid treatment and day 15. Additional assessments will be performed at month 1, 3 and 6 for those patients entering the chronic CR phase. These assessments will include at each visit: physical evaluation with neurological assessments (neurologic exam / EDSS, MSFC) and MSQLI, BMI and waist circumference to reflect the changes in body weight due to CR. Blood will be acquired on day 1, day 15 and month 3 and 6 for those patients in the CR chronic phase. This will be 15 ml of blood collected in the morning following an overnight fast. CBC, CMP and total cortisol testing will be performed by the Barnes Jewish Hospital chemistry laboratory. The rest of the blood will be processed within one hour in the investigators' laboratory. Serum will be aliquoted and stored at -80 ⁰C for future analyses (adiponectin, leptin, resistin, tumor necrosis factor-alpha and IL-6 by ELISA). The investigators will also investigate the number and function of peripheral T reg cells. T reg number will be evaluated by flow cytometry after staining fresh blood with the specific markers that identify T regs (CD4+ cells expressing high levels of CD25) and Foxp3. T reg function will be evaluated in vitro as described. Briefly, CD4+CD25high and CD4+CD25- cell populations will be isolated from peripheral blood and co-cultured at different ratios in the presence of anti cluster differentiation (CD) 3 antibodies which stimulate CD4+CD25- cell proliferation. CD4+CD25- proliferation is inhibited differentially based on the proportion of T reg cells in culture. Proliferation of CD4+CD25- cells and cytokine levels in the culture supernatants will reflect T reg suppressive capacities.

A stool sample will also be collected at baseline, day 15, month 3 and 6. These samples will be analyzed to study effects of CR on gut microbiota.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be diagnosed with relapsing MS.
* Participants must be 18 - 60 years old.
* Participants will need to be experiencing a relapse as identified by their neurologist.
* Participants must have body mass index (BMI) of 23 or higher.
* Participants must not have other ongoing diseases in other systems.

Exclusion Criteria:

* History of any chronic disease process (excluding MS) that could interfere with interpretation of results.
* Use of insulin pumps or insulin injections for diabetes.
* Use of drugs like Warfarin or Coumadin that need to monitor the intake of vegetables containing high levels of vitamin K.
* Patients that are required by a physician to follow a special diet or food restriction (diabetic, gastric bypass, soft/pureed food, etc.)
* Alcoholism, psychiatric problems, life situations that would interfere with study participation and compliance.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2014-02; Primary Completion 2016-12 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Blood biomarkers | After two weeks, 3 and 6 months
  Serum levels of: adipokines (leptin, adiponectin and resistin)
Blood biomarkers | After two weeks, 3 and 6 months
  Pro-inflammatory cytokines (IL-6, TNFalpha),
Blood biomarker | After two weeks, 3 and 6 months
  cortisol
Blood biomarker | After two weeks, 3 and 6 months
  T regulatory cell number and in vitro function

SECONDARY OUTCOMES:
Clinical - Disability on the Expanded Disability Status Scale (EDSS) | Two weeks, 3 and 6 months
  Specifically we will assess at the different time points changes in the Standardized neurologic exam called EDSS which assess clinically disability in patients with MS.
Clinical-Ambulation, hand and cognitive functions on the Multiple Sclerosis Functional Composite (MSFC) scale | Two weeks, 3 and 6 months
  The MSFC is a three-part, standardized, quantitative, assessment instrument for use in clinical studies, particularly clinical trials, of MS. (Cutter et al, 1999).
Clinical - Cognitive functions using the Symbol Digit Modality Test (SDMT). | Two weeks, 3 and 6 months
  The SDMT is a simple test to assess cognitive functions over time and assess response to treatment.
Clinical - Quality of life on the Multiple Sclerosis Quality of Life Inventory (MSQLI). | Two weeks, 3 and 6 months
  The MSQLI is a questionnaire to assess quality of life in MS patients.
Gut microbiome changes ( stool sample ) | Two weeks, 3 and 6 months
  A stool sample will be collected to assess the effect of the diet on the gut microbiome.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Piccio, MD, PhD, Principal Investigator — Washington University School of Medicine; Anne H Cross, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St Louis, St Louis, Missouri, United States

REFERENCES:
- [Background] Piccio L, Cantoni C, Henderson JG, Hawiger D, Ramsbottom M, Mikesell R, Ryu J, Hsieh CS, Cremasco V, Haynes W, Dong LQ, Chan L, Galimberti D, Cross AH. Lack of adiponectin leads to increased lymphocyte activation and increased disease severity in a mouse model of multiple sclerosis. Eur J Immunol. 2013 Aug;43(8):2089-100. doi: 10.1002/eji.201242836. Epub 2013 Jun 7. PMID 23640763
- [Background] Piccio L, Stark JL, Cross AH. Chronic calorie restriction attenuates experimental autoimmune encephalomyelitis. J Leukoc Biol. 2008 Oct;84(4):940-8. doi: 10.1189/jlb.0208133. Epub 2008 Aug 4. PMID 18678605
- [Derived] Allaf M, Elghazaly H, Mohamed OG, Fareen MFK, Zaman S, Salmasi AM, Tsilidis K, Dehghan A. Intermittent fasting for the prevention of cardiovascular disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013496. doi: 10.1002/14651858.CD013496.pub2. PMID 33512717
- [Derived] Cignarella F, Cantoni C, Ghezzi L, Salter A, Dorsett Y, Chen L, Phillips D, Weinstock GM, Fontana L, Cross AH, Zhou Y, Piccio L. Intermittent Fasting Confers Protection in CNS Autoimmunity by Altering the Gut Microbiota. Cell Metab. 2018 Jun 5;27(6):1222-1235.e6. doi: 10.1016/j.cmet.2018.05.006. PMID 29874567